CLINICAL TRIAL: NCT04523298
Title: Use of Non-ablative Vaginal Erbium YAG Laser for the Treatment of Prolapse: a Randomized Controlled Clinical Trial
Brief Title: Use of Non-ablative Vaginal Erbium YAG Laser for the Treatment of Prolapse
Acronym: VELPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Jan Deprest, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64093
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Prolapse
Keywords: laser; pelvic floor treatment
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental)
  Interventions: Procedure: Non-ablative vaginal Erbium YAG laser treatment
- PFE (Active Comparator)
  Interventions: Other: Pelvic floor exercises (PFE)

INTERVENTIONS:
Procedure: Non-ablative vaginal Erbium YAG laser treatment — There are 3 visits where vaginal application of laser will be performed, with a 4-weeks interval. If needed, 3 extra laser applications can be added to the treatment (ie. with a maximum of 6 applications). Each application lasts around 15 minutes. The vaginal laser procedure will be performed in an outpatient setting, not requiring any specific preparation, analgesia or anesthesia, by one of two experienced operators.
  Laser therapy is performed using a 2940 nm VEL (SP Spectro, Fotona, Slovenia(24)) with SMOOTH mode setting, which enables non-ablative, thermal-only operation(25). The parameters are selected based on extensive preclinical and clinical studies(26,27,28).
  Each laser treatment session consists of a full vaginal canal irradiation (using a 360° circular adapter), followed by additional irradiation of the prolapsed anterior wall (using a 90° angular adaptor) and concluded with irradiation of the vestibule area.
  Arms: Laser
Other: Pelvic floor exercises (PFE) — Standard PFE in Belgium are 9 sessions with a pelvic floor physiotherapist of choice, which can be extended by another 9 sessions, if clinically indicated. There are different strategies, though that will be on discretion of the physiotherapist. We will register the type of physiotherapy (standard (PFMT) versus assisted pelvic floor muscles training (APFMT)), number of completed sessions and duration of therapy. What is exactly done by the patient is registered as a variable.
  Arms: PFE

SUMMARY:
This is a single center, investigator initiated study, sponsored by the UZ Leuven, Leuven, Belgium; comparing laser treatment to pelvic floor exercises (PFE).

Women with symptomatic prolapse (grade II-IV) who seek for a conservative treatment, with no history of previous POP-surgery will be randomised to either the laser-arm or the PFE-arm.

There are 3 visits where vaginal application of laser will be performed, with a 4-weeks interval. Each application lasts around 15 minutes. The vaginal laser procedure will be performed in an outpatient setting, not requiring any specific preparation, analgesia or anesthesia, by one of two experienced operators.

The primary objective is to evaluate the effects of VEL treatment for reduction of prolapse symptoms and as a secondary outcome objective measurements. These endpoints are in line with the recommendations by Durnea et al., as being the most relevant and patient centered outcomes.

The second goals are to register adverse events and to determine for how long the effects of laser are sustained, with a maximum of two years. To do so, the investigators will measure long term satisfaction with, and the longevity of the effect (measured by the need for repeat or alternative therapy) of laser therapy.

Duration of follow-up per patient: max 27 months

ELIGIBILITY:
Inclusion Criteria:

* The presence of POP symptoms
* Diagnosis of cystocele or rectocele of grade II to IV according to the POP-Q system, leading the prolapse (i.e. C ≤ Ba/Bp)
* Voluntary informed consent

Exclusion Criteria:

* Symptoms or anatomical evidence for intussusception / rectal prolapse
* Leading descent of the middle compartment (C > Ba/Bp)
* Grade IV prolapse
* Previous POP surgery
* Pregnancy or <12 months postpartum
* Vaginal bleeding, injuries or infection in the treated area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-08 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the subjective improvement of POP symptoms, assessed by the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6). | 6 months after last treatment
  Participants have to answer 6 questions concerning POP symptoms with a response scale from 0 to 4 (not present (=0), not at all (=1), somewhat (=2), moderately (=3), quite a bit (=4)). The score (range 0 to 100) is then obtained by multiplying the mean value of all of the answered items by 25. Missing items are dealt with by using the mean from answered items only. Higher scores indicate more distress. This questionnaire is available and validated in English, Dutch and French. Success is defined as a reduction in scores of at least 25% compared with baseline.

SECONDARY OUTCOMES:
Assessment of the anatomical success rate by means of the POP-Q system | At every visit (ie. week 4, 8 and 12, optional: 16, 20 and 24 weeks), 6, 12 and 24 months after end of treatment
  Anatomical success is defined as POP-Q = grade 0 (no prolapse) or grade I (leading edge < -1cm)
Assessment of the rate of patient satisfaction by means of the Patient Global Impression of Improvement (PGI) | At every visit (ie. week 4, 8 and 12, optional: 16, 20 and 24 weeks), 6, 12 and 24 months after end of treatment
  a 5-point Likert scale (1=much worse, 2=worse, 3=same, 4=better, 5=much better)
Assessment of the degree of discomfort of the treatment procedure by the patient | At every visit (ie. week 4, 8 and 12, optional: 16, 20 and 24 weeks), 6, 12 and 24 months after end of treatment
  VAS-score (Visual Analogue Scale: 0-10cm, continuous scale); the higher the score, the higher the discomfort
Assessment of the longevity of the effect of laser therapy | At every visit (ie. week 4, 8 and 12), end of treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  Measured by the need for repeating the same, or initiating an alternative therapy
Assessment of sexual function, by means of the Pelvic Organ prolapse/Urinary Incontinence Sexual Questionnaire IUGA revised (PISQ-IR) | At every visit (ie. week 4, 8 and 12, optional: 16, 20 and 24 weeks), 6, 12 and 24 months after end of treatment
  The PISQ-IR is a questionnaire with twenty questions. Q1 is a question to divide the patients based on sexual activity. Not sexually active (NSA) women are referred to Q2-Q6. Sexually active (SA) women are asked to fill out Q7-Q20. The questionnaire for NSA women consists of five questions or 12 items. A higher score refers to a higher impact of PFD on sexual functioning. The questionnaire for SA women consists of 14 questions wherein women with a partner have to fill out all 14, being 22 items. Women without partner can skip questions 13 and 14, filling out 19 items. A lower score refers to a lower impact of PFD on sexual functioning. This questionnaire is available and validated in English, Dutch and French.
Assessment of urinary symptoms by means of the Urogenital Distress Inventory (UDI-6) | At every visit (ie. week 4, 8 and 12, optional: 16, 20 and 24 weeks), 6, 12 and 24 months after end of treatment
  The final UDI-6 score is calculated by adding all scores as explained in the above, and dividing the result to 6 to obtain a mean value which is in turn multiplied by 25 to obtain the scale score. The score varies from 0 to 100. The basic interpretation of the score is that the higher the score, the higher the disability. This questionnaire is available and validated in English, Dutch and French.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page AS, Borowski E, Bauters E, Housmans S, Van der Aa F, Deprest J. Vaginal erbium laser versus pelvic floor exercises for the treatment of pelvic organ prolapse: A randomised controlled trial. Eur J Obstet Gynecol Reprod Biol. 2024 Dec;303:165-170. doi: 10.1016/j.ejogrb.2024.10.042. Epub 2024 Oct 26. PMID 39488138